CLINICAL TRIAL: NCT07392489
Title: Decreasing Harms and Improving Child Health: An Intervention to Reduce Inappropriate Use of Antipsychotics and Polypharmacy
Brief Title: Decreasing Harms and Improving Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glyn Jones-Elwyn (Other)
Collaborators: Charles H. Hood Foundation (Other); Dartmouth-Hitchcock Medical Center (Other); Cayuga County Community Mental Health Center (Unknown); Clinton County Mental Health & Addiction Services (Unknown)
Responsible Party: Sponsor-Investigator, Glyn Jones-Elwyn, Professor, Trustees of Dartmouth College
Organization: Trustees of Dartmouth College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-10-216
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Psychotropic Drugs; Psychiatric Drugs; Children; Shared Decision Making; Patient Decision Aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AWARE Medication Review (Experimental): All eligible participants and their parent/caregiver take part in the AWARE intervention - a shared decision making comprehensive medication review with the participant's clinician.
  Interventions: Behavioral: AWARE Shared Decision Making Medication Review

INTERVENTIONS:
Behavioral: AWARE Shared Decision Making Medication Review — Participants, caregivers and clinicians use a shared decision making approach supported by a patient decision aid and smartphone app to review the youth's medications. This review includes discussing the original reason for the medication, how helpful the medication is, whether the youth has any side effects, the balance of side effects with effectiveness, and whether the medication is still needed. After reviewing all medications, a shared decision is made about whether to keep all medications the same or to attempt to deprescribe one of them. If the choice is to deprescribe, intervention includes a detailed, structured deprescribing protocol to support the prescribing clinician.

SUMMARY:
The investigators are doing this study because they know from research and talking with caregivers that kids can be on a bunch of medications, and it's hard to keep track of what the medications are for and whether or not they are helping.

The other thing the investigators know is that some medications have very few side effects while others have many side effects, some of which can cause real health problems (severe weight gain, diabetes). Once someone is on a medication, they often just keep taking it without thinking much about whether they still need it.

the investigators are doing this study to look at the process of reviewing medications with the help of a handout that shows basic information about the most common types of medications, making a decision about keeping medications the same or lowering one, and following people to see how it goes.

If the caregiver and youth decide to lower a medication, the investigators have created a structured process for their child's prescriber to do this slowly and safely.

Slowly means kids are not likely to have any bad reactions. This process can be used to just lower the dose of a medication or to stop it altogether.

This is called the AWARE intervention and it has 2 parts:

1. Medication review using the handout & making a decision
2. Prescribers' guide about lowering meds slowly for those who choose to do this The caregivers/youth do not have to lower a medication to be in the study.

DETAILED DESCRIPTION:
Prescriptions to children for antipsychotic medications and polypharmacy have steeply increased in recent years. Parents, schools, and clinicians may hold unrealistic expectations for these medications and desire quick relief, but do not attend to the concerning side effects or long-term morbidities. In children, the majority (75%) of antipsychotic use and 100% of polypharmacy (three or more psychiatric medications at the same time), is off-label, or not approved by the FDA for the purpose. These practices are risky, commonly leading to side effects like substantial weight gain, metabolic abnormalities, neurocognitive impairments, sedation, tremor, somnolence, and restlessness. Parents are often unaware of the risks and seldom feel fully included in decisions to use these medications. Government agencies, regulatory bodies, and media outlets have voiced significant concerns over the increased use of these medications. Clinicians and parents are interested in reducing or stopping these medications (deprescribing), but one stated barrier is the lack of guidance on how to safely deprescribe.

To address this gap, our team has developed the AWARE intervention, which incorporates two tools: 1) a patient-facing decision aid called an Option GridTM that guides both clinicians and patients/parents through a shared decision-making process about mental health treatment options; and 2) a structured protocol that provides detailed, evidence-based guidance on how to deprescribe (e.g., dose reduction rates, monitoring, safety planning) psychotropic medications in youth receiving either an off-label antipsychotic medication and/or three or more psychiatric medications concurrently. The proposed study will refine the intervention and evaluate it with 40 children receiving off-label antipsychotics or polypharmacy in two outpatient mental health clinics in the northeast.

ELIGIBILITY:
Inclusion Criteria:

* Youth will be aged 6-17 years;
* They will have been prescribed an off-label antipsychotic or polypharmacy (3 or more medications) for 3 months and be stable for 3 months (i.e. no hospitalizations or residential care).
* The parents or legal guardians of eligible children will be aged 18 years or older and capable of providing informed consent.

Exclusion Criteria:

* Children with an acute clinical or medical crisis, or a major substance use disorder will not be eligible.
* Children using an antipsychotic who have a diagnosis of psychotic disorder, bipolar affective disorder, autism spectrum disorder, or Tourette's disorder will not be eligible, as FDA approval exists for these situations.
* Youth who are pregnant will not be eligible.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | Baseline through 30-week follow-up
  The investigators measured feasibility by examining the number of people who were approached, enrolled, and completed data collection. The investigators also included the number of enrolled participants who activated their smartphone app account and accessed various sections/resources in the app.

SECONDARY OUTCOMES:
Number of medications (baseline) | Baseline
  The dose of each psychotropic medication the participant was taking was extracted from the electronic medical record and a simple count of medications was calculated. This served as the basis for measuring dose-weighted medications at 18- and 30-week follow-up.
Dose-weighted number of medications (follow-ups) | 18- and 30-week follow-up
  The investigators calculated dose-weighted medications instead of a simple medication count to reflect reductions in dose (as well as discontinuation of medications). The number of dose-weighted medications at each follow-up point was calculated as a sum of the proportion of the current daily dose of each medication compared to the sum of the baseline daily doses of those medications. For example, if a participant was taking 100 mgs of trazodone and 25 mgs of zoloft daily at baseline and 50 mgs of trazodone and 25 mgs of zoloft daily at 18-week follow-up, the dose-weighted number of medications at follow-up would be 1.5 (whereas a straight count of medications at follow-up would be 2).
Medication-related reactions | At each clinical visit (weeks 4-18)
  To facilitate data collection in this routine community setting, the investigators created the Medication Reactions Checklist (MRC), which categorizes medication reactions by body system instead of medication class. It includes all of the side effects assessed by the Psychotropic Medication Monitoring Checklist (PMMC), which is a widely-used research tool. Clinicians completed the MRC during clinic visits based on feedback gathered from the participant and caregiver.
Study-related adverse events | Ongoing monitoring throughout study participation (baseline through 30-week follow-up)
  Events meeting the NIH definition of adverse events and serious adverse events that were deemed not likely to be study related.
Columbia Impairment Scales, Parent Version (CIS-P) | Baseline, 18-, and 30-week follow-up
  The Columbia Impairment Scales, Parent Version (CIS-P) is a 13-item survey completed by the caregiver or parent that measures child functioning in four specific areas: relations with family members, relations with peers, academic or occupational functioning, and involvement in activities or interests. The scale is a 0-4 Likert scale, totals ranging from 0-52, where higher scores mean higher impairment.
Columbia Impairment Scales, Youth Version (CIS-Y) | Baseline, 18-, and 30-week follow-up
  The Columbia Impairment Scales, Youth Version (CIS-Y) is a 13-item survey completed by the caregiver or parent that measures child functioning in four specific areas: relations with family members, relations with peers, academic or occupational functioning, and involvement in activities or interests. The scale is a 0-4 Likert scale, totals ranging from 0-52, where higher scores mean higher impairment.
Modified Overt Aggression Scale (MOAS) | Baseline, 18-, and 30-week follow-up
  The Modified Overt Aggression Scale (MOAS) is a 4-item caregiver-completed measure used to capture the frequency of verbal, property-related, physical, and self-directed aggressive behaviors. Each category is scored from 0 to 4 and multiplied by weights to calculate a total weighted score ranging from 0 to 100. Higher scores demonstrate higher aggression.
Clinical Global Impression Scales - Severity (CGI-S) | Baseline, 18-, and 30-week follow-up
  The Clinical Global Impression Scales - Severity (CGI-S) is a single-item, clinician rated measure of the extent of impairment caused by mental illness symptoms that is widely utilized in pediatric clinical trials and clinical settings. It is a 7-point rating used by clinicians to assess a patient's current mental health severity (1 = normal; 7 = most severely ill).
Clinical Global Impression Scales - Improvement (CGI-I) | Baseline, 18-, and 30-week follow-up
  The Clinical Global Impression Scales - Improvement (CGI-I) is a single-item, clinician rated measure of the degree of improvement in mental illness symptoms compared to a previous assessment point, with 1 being "very much improved" and 7 being "very much worse." Like the CGI-S, it is widely utilized in pediatric clinical trials and clinical settings.

OTHER OUTCOMES:
Deprescribing choice | ~4 weeks post-baseline
  After the comprehensive medication review, participants and caregivers together with the clinician decided whether or not to try to deprescribe one of the medications. This was defined as Yes/No (decided to deprescribe/decided not to deprescribe). The investigators conceptualized this as a process outcome.
Modified Perceived Involvement in Care Scale (M-PICS) | Baseline, 18-, and 30-week follow-up
  The Modified Perceived Involvement in Care Scale (M-PICS) is a 20-item scale that measures the extent to which caregivers felt involved in clinical decisions regarding their child's care. It is scored on a 5-point Likert questionnaire (1=Never, 5=Always), where higher scores demonstrate higher involvement in care. Scores range from 20 to 100. The investigators conceptualized this as a process outcome.
CollaboRATE | -4, -8, and -12 weeks
  CollaboRATE is a caregiver-completed measure of perceived level of shared decision-making, and is a validated patient-reported experience measure that has been endorsed by the National Quality Forum. CollaboRATE contains 3 items rated on a 10-point anchored scale, with 0 indicating "No effort was made" and 9 indicating "Every effort was made." The investigators conceptualized this as a process outcome.
Weekly health functioning | during intervention (weeks 4-18)
  The investigators created a weekly health functioning measure, a health check-in rating scale to track general functioning during the study. This was scored on a 5-point scale with the response options of not at all affected, mildly affected, moderately affected, severely affected, or extremely affected. The smartphone app sent weekly prompts to caregivers to rate how much their youth had been affected in the areas of mood, behavior, sleep, ability to wake up/stay awake in the morning, ability to stay alert throughout the day, and appetite. The investigators conceptualized this as a process outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Elwyn, MD, PhD, MSc, Principal Investigator — The Dartmouth Institute for Health Policy & Clinical Practice, Geisel School of Medicine at Dartmouth
Locations (4):
- United States (4):
  - Dartmouth College, Hanover, New Hampshire
  - Dartmouth Health, Lebanon, New Hampshire
  - Cayuga County Community Mental Health Center, Auburn, New York
  - Clinton County Mental Health & Addiction Services, Plattsburgh, New York

IPD SHARING:
Plan to Share IPD: No
We do not have consent from participants to share their data.